CLINICAL TRIAL: NCT04185064
Title: Randomized-Controlled Trial and Evaluation Cohort Study of Patients Using a Cryopneumatic Device After Open or Arthroscopic Shoulder Surgeries
Brief Title: Cryopneumatic Device After Shoulder Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Encore Research Inc. (Industry)
Collaborators: CoolSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GR_001
Record Dates: First submitted 2019-11-30; First posted 2019-12-04 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Shoulder Injuries; Shoulder Disease
MeSH Terms: conditions — Shoulder Injuries | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Cryopnematic Device (Randomized Component) (Experimental): Game Ready shoulder wrap is applied in operating room and used in recovery room for 45 mins to 1 hour. Postop Day 1 and 2: the unit will be applied by the patient or a health care provider; as cold as comfortable (34°F; adjustable to 50°F); low compression setting; 30 min on:60 min off (use the pre-set auto program); use throughout the day; use at night as needed. Postop day 3-14 and onwards: 30 min on:60 min off (use the pre-set auto program); medium compression; as cold as comfortable (34°F; adjustable to 50°F); use minimum of twice/day. This will be combined with pain management medications, range of motion, and positioning exercises.
  Interventions: Device: Game Ready ATX shoulder wrap; Game Ready GRPro 2.1
- Standard Care (Active Comparator): Ice is applied in operating room and used in recovery room for 45 mins to 1 hour. Postop Day 1 and 2: the ice will be applied by the patient or a health care provider; as cold as comfortable; 30 min on:60 min off; use throughout the day; use at night as needed. Postop day 3-14 and onwards: 30 min on:60 min off; use minimum of twice/day. The patients in the control group will receive pain management strategies as would be normally dictated by the physician/therapist. This may include the use of ice, ice packs and compression bandages, as well as pain medications, range of motion, and positioning exercises
  Interventions: Other: Standard Care
- Cryopneumatic Device (Observational Cohort) (Other): Game Ready® shoulder wrap is applied in the operating room and used in the recovery room for 45 mins to 1 hour. Postop Day 1 and 2: the unit will be applied by the patient or a health care provider; as cold as comfortable (34°F; adjustable to 50°F); low compression setting; 30 min on:60 min off (use the pre-set auto program); use throughout the day; use at night as needed. Postop day 3-14 and onwards: 30 min on:60 min off (use the pre-set auto program); medium compression; as cold as comfortable (34°F; adjustable to 50°F); use minimum of twice/day. This will be combined with pain management medications, range of motion, and positioning exercises
  Interventions: Device: Game Ready ATX shoulder wrap; Game Ready GRPro 2.1

INTERVENTIONS:
Device: Game Ready ATX shoulder wrap; Game Ready GRPro 2.1 — the Game Ready ATX shoulder wrap that is anatomically engineered for the shoulder joint. The wrap is connected to the Game Ready GRPro 2.1 system enabling the integrated delivery of continuous cold and intermittent pneumatic compression therapy to the shoulder joint and surrounding soft tissues.
  Arms: Cryopnematic Device (Randomized Component); Cryopneumatic Device (Observational Cohort)
Other: Standard Care — Participants will undergo post-surgical cryotherapy using the treating surgeons preferred method of cryotherapy, which can include rest, ice, and compression using standard ice packs or bag of ice, a cryocuff, or other such device.
  Arms: Standard Care

SUMMARY:
This study randomize patients to receive either a cryopneumatic device or standard care (ice and ice packs) following open or arthroscopic shoulder surgeries. The primary objective is to determine the impact of the cryopneumatic device on post-surgery pain management, while secondary objectives are to detemine the effect on pain, patient eperience, quality of life, narcotic consumption and time to stop narcotic usage. Patients who do not wish to participate in the randomized portion of the trial will be invited to participate in an observational cohort who will all receive the cryopneumatic device. Patients who wish to enter this cohort will not have the device provided to them for free, and will either use their insurance or pay for the device, in order to determine if patients who pay demonstrate different outcomes from the patients receiving the device for free in the RCT.

ELIGIBILITY:
Inclusion Criteria:

1. men or women aged 18 years and older;
2. undergoing a unilateral primary or revision shoulder surgery (total shoulder replacement or arthroscopic surgery [rotator cuff repair, subacromial decompression, Bankart repair, Latarjet repair, debridement]).

Exclusion Criteria:

1. patients undergoing bilateral surgery;
2. patients who are pregnant or nursing;
3. patients that do not believe they can comply with the study protocol;
4. patients generally unfit for surgery;
5. patients with specific treatment preferences;
6. patients who are unable to complete questionnaires due to language barriers, decreased mental capacity, neuro-psychological problems;
7. social factors precluding follow-up; 8) inability or unwillingness to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 12 weeks
  The NPRS measures pain severity on an 11-item scale (0 to 10). The patients will be asked to choose a number from 0 to 10 that best describes their current pain. 0 would mean "no pain" and 10 would mean "worst possible pain".

SECONDARY OUTCOMES:
Narcotic Consumption | 12 weeks
  Narcotic usage will be measured based on the number of narcotics consumed during the study period and the time to cease narcotic use. Details of administration will be collected and recorded on the Medication Log CRF.
European Quality of Life measure (EQ-5D) | 12 weeks
  The European Quality of Life measure EQ-5D comprises 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) which are used to calculate a health status score from 0 (worst health) to 1 (best health). The EQ-5D also has a 0 (worst health) to 1 (best health) visual analog scale component.
Net Promoter Score | 12 weeks
  Patient experience will be measured using the Net Promoter Score. Patients will rate their experience on a simple 0 (worst) to 10 (best) scale. Responses are classified into 3 groups (promotors, passives, and distractors). The Net Promoter Score is the percentage of promoters minus the percentage of detractors.
Number of patients with adverse events; number of adverse events | 12 weeks
  All adverse events will be monitored and recorded on the Adverse Event CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Moin Khan, FRCSC, Principal Investigator — St. Joseph's Healthcare; McMaster University
Locations (5):
- Canada (5):
  - Brantford General Hospital, Brantford, Ontario
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Georgetown Hospital, Georgetown, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Oakville Trafalgar Hospital, Oakville, Ontario

IPD SHARING:
Plan to Share IPD: No
IPD will nto be shared.

REFERENCES:
- [Derived] Khan M, Phillips SA, Mathew P, Venkateswaran V, Haverstock J, Dagher D, Yardley D, Dick D, Bhandari M. Cryo-Pneumatic Compression Results in a Significant Decrease in Opioid Consumption After Shoulder Surgery: A Multicenter Randomized Controlled Trial. Am J Sports Med. 2024 Sep;52(11):2860-2865. doi: 10.1177/03635465241270138. Epub 2024 Aug 21. PMID 39165152